CLINICAL TRIAL: NCT06046690
Title: Comparison of the Effects of Inspiratory Muscle Training with Trigger System Modification and External Device in Mechanically Ventilated Patients
Brief Title: Comparison of the Effects of Inspiratory Muscle Training Methods in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other); SB Goztepe Prof Suleyman Yalcin City Hospital (Unknown)
Responsible Party: Principal Investigator, Mehmet Burak Uyaroğlu, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SaglikBilimleriUni
Record Dates: First submitted 2023-08-22; First posted 2023-09-21 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-01

CONDITIONS: Mechanical Ventilation; Intensive Care Units
Keywords: İnspiratory muscle training; intensive care; rehabilitation; mechanical ventilation
MeSH Terms: interventions — External Fixators

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MV Modification Group (Experimental): Participant in this group will be applied inspiratory muscle training with trigger system modification in addition to conventional chest physiotherapy consisting of respiratory control, diaphragmatic breathing, costal expansion exercises, postural drainage, effective coughing, in-bed ROM exercises and mobilization, twice a day until the day of extubation.
  Interventions: Device: Mechanical Ventilation Device
- External Device Group (Experimental): Participant in this group will be applied inspiratory muscle training with Inspiratory Muscle Training (IMT) device in addition to conventional chest physiotherapy consisting of respiratory control, diaphragmatic breathing, costal expansion exercises, postural drainage, effective coughing, in-bed ROM exercises and mobilization, twice a day until the day of extubation.
  Interventions: Device: External Device

INTERVENTIONS:
Device: Mechanical Ventilation Device — During the first week of training, ventilator trigger sensitivity will be initiated at 20% of the patient's baseline MIP (NIF). Patients will train for 5 minutes twice a day for the first days. As the training progresses, the triggering sensitivity will be gradually increased to 30% and 40% of the initial MIP and the duration will be increased up to 30 minutes. During the training sessions, participants will be elevated to a position similar to the Semi-Fowler position at an angle of approximately 45°. Vital signs will be monitored regularly.
  In addition, conventional chest physiotherapy consisting of respiratory control, diaphragmatic breathing, costal expansion exercises, postural drainage, effective coughing, in-bed ROM exercises and mobilization will be applied twice daily.
  Arms: MV Modification Group
Device: External Device — The IMT (Inspiratory Muscle Training) with device will commence at 20% of the value obtained from the NIF (Negative Inspiratory Force) measurement or the lowest pressure setting, depending on the patient's tolerance. The duration and intensity will be gradually increased. Once the participants are disconnected from the mechanical ventilator, the IMT device will be connected to the T-tube via a catheter mount with a Catheter Mount. Patients will be instructed to breathe against the resistance set on the IMT device. After completing 8 repetitions, the patient will be allowed to rest for a few minutes. This routine will be repeated for a total of 3 sets of 8 repetitions.
  In addition, conventional chest physiotherapy consisting of respiratory control, diaphragmatic breathing, costal expansion exercises, postural drainage, effective coughing, in-bed ROM exercises and mobilization will be applied twice daily.
  Arms: External Device Group

SUMMARY:
Inspiratory Muscle Training(IMT) increases the strength and endurance of the inspiratory muscles, exercise capacity, quality of life and reduces the perception of dyspnea. It has been reported in the literature that it also has an effect on mechanical ventilated patients in the intensive care unit. In patients on mechanical ventilation, IMT is applied with modification of trigger sensitivity and with an external device.

The aim of this study is to compare the effects of inspiratory muscle training with external device and MV modification on respiratory muscle strength and intubation time

DETAILED DESCRIPTION:
The intensive care unit (ICU) is the unit where patients with acute and life-threatening organ dysfunction or at risk are treated. Various technologies are used to support organ systems, especially the lungs, cardiovascular system, and kidneys. Mechanical ventilation (MV) device is the most important of these technologies. The device is clinically used in patients who need assistance to maintain adequate alveolar ventilation. Although MV is a life-saving intervention in respiratory failure, both short-term and longterm harmful consequences have been proven. Patients are weaned from mechanical ventilation when they begin to effective breathing on their own. However, he has persistent problems during his stay at the MV. Prolongation of the time spent on mechanical ventilation; It prolongs hospital stay and increases mortality and morbidity with many secondary pathologies ranging from pneumonia to polyneuropathy to delirium. As a result of all these, MV of the patient may cause reused. Physiotherapy is a very important component in the treatment of ICU patients, with both short-term and long-term advantages. Respiratory physiotherapy provides positive changes in hemodynamic and respiratory physiological parameters. Chest physiotherapy methods such as various chest manipulations, chest vibration and percussion, manual hyperinflation, postural drainage and various coughing techniques can be applied together or separately to prevent pulmonary complications in ICU patients. Techniques are used in mechanically ventilated patients to maintain airway clearance, reduce work of breathing, expand lungs, and prevent complications. Inspiratory muscle training (IMT), one of the respiratory physiotherapy applications used, is a technique used to increase the strength and endurance of the diaphragm and other accessory inspiratory muscles. In the ICU, inspiratory muscle training is achieved through devices that apply resistance or load to the inspiratory muscles, or through modification of the mechanical ventilator.

The aim of this study is to compare the effects of inspiratory muscle training with external device and MV modification on respiratory muscle strength and intubation time.

This prospective study will be conducted in Goztepe Prof. Dr. Suleyman Yalcın Cıty Hospıtal Hospital, Intensive Care Unit. Thirty-eight mechanically ventilated patients will be included in the study and randomly divided into two groups. In the MV group(MV-GR)(n=19), will be applied IMT with MV modification in addition to conventional physiotherapy, while in the external device group (E-GR) (n=19), IMT will be applied with an additional external device to conventional physiotherapy. P-FIT scale will be used for evaluation criteria, maximal inspiratory pressure, rapid shallow breathing index, oxygenation index, tidal volume, minute ventilation, weaning success values and functional status.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age,
* Hemodynamically stable,
* Alert and conscious(Between -2 and +2 according to Richmond Agitation and Sedation Scale score)
* Perform at least one motor command,
* Requiring mechanical ventilation support either with continuous spontaneous ventilation(CPAP) mode or intermittent mandatory ventilation(SIMV) mode with pressure or volume control(PSV),
* Requiring oxygen ventilation ≤ 40%, Required pressure support ≤ 15 cmH2O, and PEEP ≤ 10 cmH2O,
* Having a body temperature between 36- 38 °C,
* Unable to breathe unsupported for 72 consecutive hours following the resolution of factors supporting respiratory failure,
* Having FiO2 ≤ 0.5, PaO2 > 60 mmHg, and capable of sufficient gas exchange,
* Patients deemed suitable for pulmonary physiotherapy by intensive care physicians will be included in the study.

Exclusion Criteria:

* Having an acute onset of illness,
* Impaired cooperation,
* Insufficient level of consciousness due to severe intracranial disease ,
* Having a progressive neuromuscular disease,
* Having an unstable neurological condition,
* Having a psychiatric disorder and exhibiting excessive agitation (patients with Richmond Agitation and Sedation Scale (RASS) ≥ +2),
* Having experienced any trauma to the chest wall,
* Having thoracic deformities that affect respiration,
* Using a high amount of sedative or analgesic agents,
* Participants using home mechanical ventilators prior to hospital admission.

Criteria for Study Discontinuation:

* Cardiac, pulmonary, and other conditions leading to impaired hemodynamic stability.
* Impaired cooperation, compliance, and motivation.
* Discontinuation by the intensive care physician.
* Participants will be free to withdraw from the study at their discretion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Assesment of respiratory muscle strength | It will be measured before training and before extubation.
  Negative inspiratory force (NIF) is the maximum pressure that can be generate against an occluded airway and is a marker of respiratory muscle function and strength. The Negative Inspiratory Force index (NIF) measures the patient's maximum inhalation effort after exhaling. This value is also known as the Maximum Inspiratory Pressure (MIP). Patients with a NIF < -30mbar (more negative) can in all probability be weaned successfully, while those with a NIF of up to -20mbar (less negative) will most probably prove unsuccessful and weaning is more likely to fail. The NIF is measured as a pressure against PEEP (Positive end-expiratory airway pressure).
Assesment of lung volume assessment | Measurements will be taken before and after daily exercises from the start of education until the day of extubation, an average 10 days
  While in CPAP mode, the participants will be instructed to take deep breaths and exhale for about 1 minute with Pressure Support value 10 cmH2O and PEEP 5 cmH2O. At this time, the highest inspiratory tidal volume and expiratory tidal volume in milliliters (ml) will be recorded.
Assesment of the respiratory status | It will be measured before training and before extubation.
  Rapid Shallow Breathing Index (RSBI) is calculated by dividing the respiratory rate (number of breaths) by the tidal volume (volume of air in each breath). The formula is as follows:
  RSBI = Respiratory Rate / Tidal Volume Low RSBI values indicate that the patient tolerates mechanical ventilation well and there is minimal fatigue in the respiratory muscles. High RSBI values may suggest fatigue and increased strain on ventilation.
Assesment of the oxygenation status | It will be measured before training and before extubation.
  Oxygenation Index (OI) is used to evaluate a mechanically ventilated patient's oxygenation (oxygen level) in relation to the need for respiratory support. The formula is as follows:
  OI = (Oxygen Pressure / Fraction of Inspired Oxygen) * Mean Airway Pressure Low OI values indicate good oxygenation and low requirement for respiratory support, while high OI values may indicate poor oxygenation and a greater need for respiratory assistance.
Assesment of physical status | It will be measured before training and before extubation.
  The PFIT-S is a specific assessment tool designed to measure the physical function of patients in the intensive care unit (ICU). It aims to evaluate the patient's ability to perform various physical tasks and activities during their ICU stay. The PFIT-S helps healthcare professionals assess the patient's functional status, track their progress, and guide rehabilitation interventions. It includes 4 items: amount of assistance for sit-to-stand transfers, strength for shoulder flexion, strength for knee extension, marching in place.The PFIT-s scores range from 0 (able to perform strength testing only with a maximal score of 2/5 for shoulder and knee) to 10 (performance without any difficulty)
Assesment of Mechanical ventilator parameters | Measurements will be taken before and after daily exercises from the start of education until the day of extubation, an average 10 days
  Before the training, the mechanical ventilator mode, PEEP (Positive End-Expiratory Pressure), Pressure support values in cmH2O of the participants will be recorded.
Assesment of Partial Pressure of Oxygen(PaO2) and Partial Pressure of Carbon dioxide(PaCO2) in Arterial Blood | Measurements will be taken before and after daily exercises from the start of education until the day of extubation, an average 10 days
  PaO2(mmHg) and PaCO2(mmHg) in the blood represents the respective concentrations of these gases dissolved in the blood plasma. These values are crucial indicators of respiratory function and metabolic balance within the body. Monitoring these partial pressures is fundamental in assessing respiratory efficiency and guiding appropriate medical interventions for patients with various health conditions.
Assesment Concentration of Bicarbonate(HCO3) in Arterial Blood | Measurements will be taken before and after daily exercises from the start of education until the day of extubation, an average 10 days
  HCO3 (meq/L) aids in discerning the extent or seriousness of anomalies, distinguishing between acute and chronic abnormalities, and identifying whether the primary condition is metabolic or respiratory in nature. Automated blood gas analyzers are used to analyze blood gas samples and define HCO3 values
Assesment pH values | Measurements will be taken before and after daily exercises from the start of education until the day of extubation, an average 10 days
  A pH of 7.37 is classified as acidosis, while a pH of 7.42 is categorized as alkalemia. Automated blood gas analyzers are used to analyze blood gas samples and define pH values
Assesment of Minute Ventilation | Measurements will be taken before and after daily exercises from the start of education until the day of extubation, an average 10 days
  While in CPAP mode, the participants will be instructed to take deep breaths and exhale for about 1 minute with Pressure Support value 10 cmH2O and PEEP 5 cmH2O. The highest minute ventilation in liters per minute (l/min), will be recorded
Assesment Fraction of Inspired Oxygen(FiO2) | Measurements will be taken before and after daily exercises from the start of education until the day of extubation, an average 10 days
  FiO2, refers to the concentration of oxygen in the air being delivered to a patient during mechanical ventilated. It plays a crurial role in managing patients with respiratory conditions, as it helps healthcare professionals adjust oxygen therapy to maintain adequate oxygenation and prevent complications like hypoxia or oxygen toxicity. Precise monitoring and adjustment of FiO2 levels are essential in optimizing patient care and outcomes in clinical settings.Before the training FiO2 in % of the participants will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Kocoglu, Prof.Dr., Study Chair — Goztepe Prof Dr Suleyman Yalcın City Hospital; Esra Pehlivan, Ass.Prof., Principal Investigator — Saglik Bilimleri Universitesi; Mehmet Burak Uyaroglu, PT,PhD(c), Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)